CLINICAL TRIAL: NCT05950399
Title: Evaluating Changes in Cardiac Function During Stress Echocardiography for the Identification of Chemotherapy Induced Cardiotoxicity in Cancer Patients at Risk of Developing Heart Failure
Brief Title: Stress Echocardiography to Identify Chemotherapy Induced Cardiotoxicity in Cancer Patients With Heart Failure Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15-002855; NCI-2022-10806 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-002855 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (resting and/or stress echocardiography) (Experimental): Patients choose to undergo either a resting echocardiography performed before and after delivery of a cancer therapeutic agent and months 3, 6, 9 and 12 or up to 5 low intensity stress echocardiography over 25 minutes performed depending on where they are at in the course of their cancer therapy and/or cardiac rehabilitation program at baseline and/or months 3, 6, 9 and 12 after starting cancer therapy.
  Interventions: Procedure: Echocardiography; Other: Electronic Health Record Review; Other: Questionnaire Administration; Procedure: Stress Echocardiography
- Group II (stress echocardiography) (Active Comparator): Participants undergo low intensity stress echocardiography over 25 minutes at baseline and may undergo a second one at least 24 hours later.
  Interventions: Procedure: Stress Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Undergo resting echocardiography
  Other Names: EC
  Arms: Group I (resting and/or stress echocardiography)
Other: Electronic Health Record Review — Ancillary studies
  Arms: Group I (resting and/or stress echocardiography)
Other: Questionnaire Administration — Ancillary studies
  Arms: Group I (resting and/or stress echocardiography)
Procedure: Stress Echocardiography — Undergo stress echocardiography
  Other Names: Stress Echo

SUMMARY:
This clinical trial evaluates changes in cardiac (heart) function during stress echocardiography to screen for chemically induced cardiotoxicity in cancer patients at a high risk for developing heart failure. Some chemotherapeutic agents to treat certain types of cancers can induce cardiac dysfunction and heart failure. Currently there is no validated means of predicting which patients will go on to develop cardiac toxicity and heart failure following treatment with chemotherapeutic agents. Stress echocardiography is a test that uses ultrasound imaging to show how well the heart muscle is working to pump blood to the body during low intensity exercise. Stress echocardiography prior to and during cancer treatment may help doctors find cancer therapeutic related cardiac dysfunction sooner when it may be easier to treat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether changes in the following parameters of cardiac function at rest or with low intensity exercise occur following (1) treatment with cancer therapeutics or (2) cardiac rehabilitation:

Ia. 2-Dimensional (2D) and 3-dimensional (3D) left ventricular (LV) longitudinal strain and strain rate; Ib. Right ventricular (RV) longitudinal strain and strain rate; Ic. LV circumferential and radial strain and strain rate; Id. 2D and 3D wall motion; Ie. 2D and 3D volumetric left ventricular ejection fraction (LVEF); If. Mitral valve inflow velocities (E, A) and mitral annular tissue Doppler (e', a'); Ig. Tricuspid tissue velocities and tricuspid annular plane systolic excursion (TAPSE).

SECONDARY OBJECTIVES:

I. To determine whether changes after treatment with cancer therapeutics or a period of cardiac rehabilitation in any of the aforementioned parameters of cardiac function with low intensity exercise:

Ia. Occur before changes in resting strain or resting LVEF; Ib. Predict future reductions in LVEF (cardiotoxicity) or in the case of cardiac rehabilitation, prevention of LVEF decrease; Ic. Predict the development of clinical heart failure.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I (CASE): Patients choose to undergo either a resting echocardiography performed before and after delivery of a cancer therapeutic agent and months 3, 6, 9 and 12 or up to 5 low intensity stress echocardiography over 25 minutes performed depending on where they are at in the course of their cancer therapy and/or cardiac rehabilitation program at baseline and/or months 3, 6, 9 and 12 after starting cancer therapy.

GROUP II (CONTROL): Participants undergo low intensity stress echocardiography over 25 minutes at baseline and may undergo a second one at least 24 hours later.

After completion of study intervention, patients in Group 1 are followed up at 2, 5, and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous diagnosis of solid organ cancers (breast, non-small cell lung, rectal, renal, hepatic cancer, metastatic melanoma, sarcoma) or hematological disease (lymphoma, leukemia, multiple myeloma, monoclonal gammopathy of undetermined significance [MGUS])
* Age >= 18 years at study enrollment
* Plan to receive, or history of having received, chemotherapy (anthracycline, alkylating agent [cyclophosphamide, ifosfamide], and/or antimicrotubule agent [docetaxel, paclitaxel]) with or without specific targeted therapies;

  * Anti-HER2 targeted therapies (trastuzumab, pertuzumab)
  * Vascular endothelial growth factor (VEGF) inhibitors (bevacizumab, sunitinib, sorafenib, pazopanib, axitinib, vandetanib)
  * Immune checkpoint inhibitors (ipilimumab, nivolumab, pembrolizumab)
* Plan to undergo conditioning chemotherapy for bone marrow transplantation (autologous/allogeneic)

Exclusion Criteria:

* Coronary artery disease
* Significant (more than mild) valvular heart disease
* Pre-existing heart failure
* Pre-existing cardiomyopathy
* Musculoskeletal or neurologic abnormality prohibiting low intensity exercise on a stationary bicycle
* Severe pulmonary disease limiting ability to perform low intensity exercise on a stationary bicycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac function with low intensity exercise in cancer patients | Baseline to 12 months
  Resting echocardiography will be performed immediately before and after patient receives cancer therapeutic treatment. Up to five sessions of low intensity stress echocardiograms will be performed during the course of the study depending on where they are in the course of cancer therapy and/or cardiac rehabilitation program at study enrollment. Patients may opt to change from low intensity echocardiogram to resting echocardiogram during the course of the study.
Changes in cardiac function with low intensity exercise in cancer patients after treatment with cancer therapeutics. | Baseline to 12 months
  Resting echocardiography will be performed immediately before and after patient receives cancer therapeutic treatment. Up to five sessions of low intensity stress echocardiograms will be performed by during the course of the study depending on where they are in the course of cancer therapy and/or cardiac rehabilitation program at study enrollment. Patients may opt to change from low intensity echocardiogram to resting echocardiogram during the course of the study. D
Changes in cardiac function with low intensity exercise in cancer patients after a period of cardiac rehabilitation. | Baseline to 12 months
  Resting echocardiography will be performed immediately before and after patient receives cancer therapeutic treatment. Up to five sessions of low intensity stress echocardiograms will be performed by during the course of the study depending on where they are in the course of cancer therapy and/or cardiac rehabilitation program at study enrollment. Patients may opt to change from low intensity echocardiogram to resting echocardiogram during the course of the study.

SECONDARY OUTCOMES:
Reductions in left ventricular ejection fraction (LVEF) | Up to 10 years
  Data will be collected from chart reviews and patient surveys. Predictors of reductions in LVEF will be assessed using linear regression and multiple linear regression analyses. A p-value < 0.05 will define significance. Cancer Therapeutics-Related Cardiac Dysfunction will be defined as per recent guidelines as a drop in LVEF of > 10% to < 53%.
Reductions in onset of clinical heart failure | Up to 10 years
  Data will be collected from chart reviews and patient surveys. Predictors of reductions in heart failure will be assessed using linear regression and multiple linear regression analyses. A p-value < 0.05 will define significance. Heart failure will be defined as a diagnosis made by one of the patients treating physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Hector R Villarraga, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials